CLINICAL TRIAL: NCT03664505
Title: Evaluation of the Product Properties of Individualized 3D-compression Garments to Treat Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, Principal Investigator, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-174
Record Dates: First submitted 2018-08-31; First posted 2018-09-10 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Burn Scar
MeSH Terms: interventions — Radionuclide Imaging

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient receives two different burn garments and does not know which one was produced based on the scan data and which one on the manual measuring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garment based on manual measurement (Active Comparator): Garment based on manual measurement is used on burn scar
  Interventions: Device: Compression garment (manual)
- Garment based on scan measurement (Experimental): Garment based on scan measurement is used on burn scar
  Interventions: Device: Compression garment (scan)

INTERVENTIONS:
Device: Compression garment (manual) — Garment based on manual measurement
  Arms: Garment based on manual measurement
Device: Compression garment (scan) — Garment based on scan measurement
  Arms: Garment based on scan measurement

SUMMARY:
Burn scars are treated with compression garments. These are produced based on manual measure data. The aim of this study is to evaluate correct fitting, wearing comfort, suitability for daily use and scar properties after using garments produced on base of measuring data from scanning in comparison to manual measured data.

DETAILED DESCRIPTION:
In plastic and reconstructive surgery, treatment of burn scars is still challenging, because excessive and hypertrophic scarring can occur. Burn garments are usually used to reduce such scarring. However, measure are taken manually by a measuring tape using interpolation. Therefore, compression garments produced on base of 3D surface imaging using a scanning system are compared to compression garments based on manually measurements regarding correct fitting, wearing comfort, suitability for daily use and scar properties.

ELIGIBILITY:
Inclusion Criteria:

* Burn scars on an arm after IIa-III. burn (1-30% surface area)
* Indication for burn garments
* Experience in using burn garments

Exclusion Criteria:

* Consume of pain killer
* Medication with cortisone or immun suppressive therapy
* Psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Fitting of the garment (on a numeric rating scale 0-10) | 3 months
  Numeric rating scale from 0 (minimum) to 10 (maximum) judged by the patient: 0 means perfect fitting, 10 means no fitting). Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Comfort of the garment (on a numeric rating scale 0-10) | 3 months
  Numeric rating scale from 0 (minimum) to 10 (maximum) judged by the patient: 0 means good wearing comfort, 10 means bad wearing comfort. Higher values represent a worse outcome.
Daily use of the garment (on a numeric rating scale 0-10) | 3 months
  Numeric rating scale from 0 (minimum) to 10 (maximum) judged by the patient: 0 means good suitability of daily use, 10 means bad suitability of daily use. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No